CLINICAL TRIAL: NCT02803606
Title: Evaluation of Risk Factors Predictive of Hypothermia in Preterm Neonates in Incubators During the First Week of Life
Acronym: PREMARISQ
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: AOL08-DR-TOURNEUX
Record Dates: First submitted 2016-06-06; First posted 2016-06-17 (Estimated); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Hypothermia
Keywords: hypothermia; routine care; preterm neonates
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- hypothermia: Preterm neonates less than 32 weeks of gestational age admitted at birth to the Neonatal Medicine unit

SUMMARY:
Preterm neonates less than 32 weeks of gestational age admitted at birth to the Neonatal Medicine unit will be included after informing the parents. Abdominal skin and peripheral (arm or leg) and incubator air temperatures and relative humidity will be obtained from data recorded by the incubator without using any additional transducer compared to standard care. Pulse and respiratory rate, blood pressure, the incidence of apnoeas and sleep organization will also be recorded from routine monitoring. A case report form and a wide-angle video recording of the infant's room will allow description of the type of care, determine the duration of care and the impact on incubator function. Data will be recorded for the first 7 days of life of the preterm neonate.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants of 25-32 weeks of gestation
* Birth in one of the two maternity hospitals of Amiens agglomeration (CGO or clinic of Europe )
* Arrived in the Neonatal Medicine unit < 2 hours of life
* Necessitated a care in an incubator

Exclusion Criteria:

* Preterm infants > 32 weeks of gestation
* Birth outside the Amiens metropolitan area
* Arrived in the Neonatal Medicine unit after 2 hours of life
* Present a malformation syndrome or severe heart disease
* Pathology requiring support within the first 7 days of life
* Apgar score < 5 to 10 minutes of life
* Need for initial management in open incubator
* Unavailability of a type of incubator " Caleo® "

Ages: 25 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm neonates less than 32 weeks of gestational age admitted at birth to the Neonatal Medicine unit
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2009-06; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Lowest abdominal skin temperature | 20 minutes

SECONDARY OUTCOMES:
The nadir for peripheral skin temperature | 20 minutes
Pulse rate | 20 minutes
Morbidity | 7 days
mortality | 7 days
respiratory rate | 20 minutes
Blood pressure | 20 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Pierre TOURNEUX, MD,PhD, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France